CLINICAL TRIAL: NCT01138995
Title: Functional Ambulation: Standard Treatment vs. Electronic Stimulation Therapy (FASTEST)Trial in Chronic Post-Stroke Subjects With Foot Drop
Brief Title: Clinical Study of the L300 Versus Ankle-foot Orthosis (AFO) on Post-Stroke Subjects With Foot Drop
Acronym: L300
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioness Inc (Industry)
Collaborators: Medidata Solutions (Industry); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-L300-0801, Rev. B
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-03

CONDITIONS: Sensorimotor Gait Disorder; Neurologic Ambulation Disorder; Gait, Drop Foot; Poststroke Hemiparesis; Post-Cerebrovascular Accident (CVA) Hemiparesis
Keywords: Poststroke/CVA hemiparesis; Drop Foot; Gait Disorders, Neurological; Gait, Drop foot
MeSH Terms: conditions — Gait Disorders, Neurologic; Stroke; Paresis; Peroneal Neuropathies; Mobility Limitation; Neurologic Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ankle-foot orthosis (AFO) Control Group (Active Comparator): The Control Group will walk with the a "usual" ankle-foot orthosis (AFO) for 30 weeks.
  Interventions: Device: Ankle-foot orthosis
- Ness L300 Treatment Group (Experimental): The Original Treatment Group will walk with the Ness L300 for 30 weeks.
  Interventions: Device: Ness L300

INTERVENTIONS:
Device: Ness L300 — The Ness L300 delivers functional electrical stimulation (FES), which improves gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
  Other Names: Leg Stimulator
  Arms: Ness L300 Treatment Group
Device: Ankle-foot orthosis — The Control Group will walk with a "usual" ankle-foot orthosis (AFO).
  Other Names: drop foot orthotic
  Arms: Ankle-foot orthosis (AFO) Control Group

SUMMARY:
The objective of this study is to determine the effectiveness of the NESS L300 (L300) in improving gait parameters, function, and quality of life among stroke subjects (greater than or equal to 3 months post stroke)with drop foot.

DETAILED DESCRIPTION:
Approximately 176 subjects with stroke that have drop foot will be enrolled from approximately 10 different sites in the United States depending on the rate of enrollment. This clinical study is proposed to show that the functional electrical stimulation (FES) delivered via the Ness L300 improves gait function, stroke-specific quality of life, and safety for persons with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Have ankle dorsiflexion range of motion greater than or equal to neutral when assessed concurrent with test stimulation in sitting and standing and demonstrate adequate ankle and knee stability during gait at the time of screening
* Have had at least one stroke of any etiology (e.g., ischemic, hemorrhagic,etc.) experienced greater than or equal to 3 months prior to study enrollment, as confirmed by independent medical records, and result in drop foot sufficient to require prior or current prescription for and/or use of an AFO
* Have adequate cognition and communication abilities for informed consent, training and instructions, use of the L300, and provide feedback, to be demonstrated by either the subjects scoring greater than or equal to 24 (out of a possible 30) on the Mini Mental State Examination, or having a competent caregiver for these purposes
* Must be 18 years or older
* Have the ability to safely walk at least 10-meters with a maximum of 1 person assist
* Have a self-selected 10-meter gait speed of less than or equal to 0.8m/s at the time of assessment
* Have inadequate dorsiflexion/limb clearance or unable to achieve normal heel strike on ambulation without AFO
* Be medically stable

Exclusion Criteria:

* Have fixed ankle contracture at greater than or equal to 5 degrees of plantar flexion in the hemiplegic leg with the knee extended
* Have excessive pain in the affected leg, as measured by a score greater than or equal to 4 on a 10-point visual analog scale
* Participation, within the past 3 months, currently, or during the course of the study in any interventional clinical studies without the Sponsor's approval
* Have a demand-type cardiac pacemaker, defibrillator, or any electrical or metallic implant
* Have a lower motor neuron disease or injury with inadequate response to stimulation
* Have significant swelling/edema in the leg extending up to the knee
* Have a history of chronic skin problems/conditions or cancerous lesion present or suspected in close proximity ot the expected site for L300 stimulation
* Are pregnant or plan on becoming pregnant in the next 45 weeks
* Have had botulinum toxin(type a or b) to the hemiplegic leg or arm within the past six weeks or plan to have botulinum toxin treatments during the course of the study
* Expectation of a significant change in the subject's spasticity medications during the course of the study for the effected leg
* Have unstable seizure disorder (average of greater or equal to 2 seizures per month)
* Have a pre-existing significant orthopedic conditions that are, a that investigator's discretion, determined as likely to limit ambulatory progress (e.g., total hip replacement [non-metallic], total knee replacement [non-metallic], limited lower extremity (LE) range of motion (ROM), rheumatoid arthritis, osteoarthritis, or other fracture or dislocation that underlies the expected site for L300 stimulation)
* Have a complete hemisensory loss ipsilateral to foot drop
* Used the L300 or other FES device for foot drop (e.g., Odstock Drop Foot System (ODFS), WalkAide by Innovation Neurotronics, etc.) for greater than or equal to 3 hours within the last 6 months prior to study enrollment
* Have major post-stroke depression (PHQ-9 greater than or equal to 10) that is not medically managed with antidepression medication and/or psychotherapy
* Currently or planning on participating in a neuro-rehabilitation physical therapy (PT) or occupational therapy (OT) program or new independent exercise programs with enrolled in the study. However, injury or a change in condition requiring PT or OT that would not affect gait outcomes maybe assessed by an off-site study committee, on a case-by-case basis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kari Dunning, PT, Ph.D, Study Chair — The Drake Center/University of Cincinnati; Michael O'Dell, MD, Study Chair — Weill Medical College of Cornell University; Patricia Kluding, PT, Ph.D., Principal Investigator — University of Kansas; Steven R. Edgley, MD, Principal Investigator — University of Utah; Kathaleen P Brady, PT, NCS, Principal Investigator — MedStar National Rehabilitation Network; Trevor Paris, MD, Principal Investigator — Brooks Rehabilitation; Jerome Stenehjem, MD, Principal Investigator — Sharp Rehabilitation Center; John Thottakara, MD, Principal Investigator — UT Southwestern; Jun Zhang, MD, Principal Investigator — St. Charles Hospital & Rehabilitation; Ziyad Ayyoub, MD, Principal Investigator — Rancho Los Amigos National Rehabilitation; Diemha Hoang, MD, Principal Investigator — Long Beach Memorial Medical Center
Locations (11):
- United States (11):
  - Rancho Los Amigos National Rehabilitation Center, Downey, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Sharp Rehabilitation Center, San Diego, California
  - National Rehabilitation Hospital, Washington D.C., District of Columbia
  - Brooks Center for Rehabilitation Studies, Jacksonville, Florida
  - Kansas University Medical Center, Kansas City, Kansas
  - Weill Cornell Medical Center, New York, New York
  - St.Charles Hospital & Rehabilitation, Port Jefferson, New York
  - The Drake Center /University of Cincinnati, Cincinnati, Ohio
  - UT Southwestern, Dallas, Texas
  - University of Utah, School of Medicine, Salt Lake City, Utah

REFERENCES:
- [Derived] Alenazi AM, Alshehri MM, Alothman S, Rucker J, Dunning K, D'Silva LJ, Kluding PM. Functional Reach, Depression Scores, and Number of Medications Are Associated With Number of Falls in People With Chronic Stroke. PM R. 2018 Aug;10(8):806-816. doi: 10.1016/j.pmrj.2017.12.005. Epub 2017 Dec 26. PMID 29288141
- [Derived] O'Dell MW, Dunning K, Kluding P, Wu SS, Feld J, Ginosian J, McBride K. Response and prediction of improvement in gait speed from functional electrical stimulation in persons with poststroke drop foot. PM R. 2014 Jul;6(7):587-601; quiz 601. doi: 10.1016/j.pmrj.2014.01.001. Epub 2014 Jan 9. PMID 24412265
- [Derived] Kluding PM, Dunning K, O'Dell MW, Wu SS, Ginosian J, Feld J, McBride K. Foot drop stimulation versus ankle foot orthosis after stroke: 30-week outcomes. Stroke. 2013 Jun;44(6):1660-9. doi: 10.1161/STROKEAHA.111.000334. Epub 2013 May 2. PMID 23640829

RESULTS

PARTICIPANT FLOW:
Groups:
- Originial Control Group: The Control Group will walk with the a "usual" ankle-foot orthosis (AFO)for 30 weeks. After 30 weeks, the Original Control Group will then be crossed over to walk with the Ness L300 for a total of 12 weeks.
  Ness L300: The Ness L300 delivers functional electrical stimulation (FES), which improves gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
  Ness L300: The Original Treatment Group will walk with the Ness L300 for 42 weeks, and the Original Control Group will walk with a "usual" ankle-foot orthosis (AFO)for 30 weeks, then be crossed over to walk with the Ness L300 for a total of 12 weeks.
- Original Treatment Group: The Original Treatment Group will walk with the Ness L300 for 42 weeks.
  Ness L300: The Ness L300 delivers functional electrical stimulation (FES), which improves gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
  Ness L300: The Original Treatment Group will walk with the Ness L300 for 42 weeks, and the Original Control Group will walk with a "usual" ankle-foot orthosis (AFO)for 30 weeks, then be crossed over to walk with the Ness L300 for a total of 12 weeks.
Period: Overall Study
Arm/Group | Originial Control Group | Original Treatment Group
Started | 98 | 99
Completed | 88 | 74
Not Completed | 10 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Originial Control Group | Original Treatment Group | Total
Number analyzed (Participants) | 98 | 99 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.9) | 60.7 (12.2) | 61.1 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 48 | 79
  Male | 67 | 51 | 118
Region of Enrollment [Number; unit: participants]
  United States | 98 | 99 | 197

OUTCOME MEASURES:

1. Primary Outcome: Ten Meter Walk Test (10mWT)
Description: Determine gait velocity during a 10 meter walk test for subjects using the L300 versus subjects using a standard "usual" ankle-foot orthosis (AFO). Long term device effect at comfortable gait speed in m/s. Walk test results at 30 weeks will be compared to baseline speed. The mean difference (improvement) between baseline and week 30 will be presented by study arm.
Time Frame: Week 30
Population: Intent to treat analysis of 197 (98 Control and 99 Treatment) randomized subjects.
Measure: Mean (Standard Deviation); unit: meters per second (m/s)
Groups:
- Originial Control Group: The Control Group will walk with the a "usual" ankle-foot orthosis (AFO)for 30 weeks.
- Original Treatment Group: The Original Treatment Group will walk with the Ness L300 for 30 weeks.
  The Ness L300 delivers functional electrical stimulation (FES), which improves gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
Arm/Group | Originial Control Group | Original Treatment Group
Number analyzed (Participants) | 98 | 99
meters per second (m/s) | 0.15 (0.14) | 0.14 (0.16)
Statistical Analysis 1: Comparison: Originial Control Group vs Original Treatment Group; Test type: Superiority or Other; p = 0.75, Fisher's combination test; Between group difference for entire sample

2. Secondary Outcome: Berg Balance Scale (BBS) Score
Description: Clinical measurement of balance was recorded using the Berg Balance Scale which is a highly reliable and valid test used among persons with stroke. This Scale consists of 14 items/tasks of increasing difficulty graded on a five-point ordinal scale of zero to four where zero = participant is unable to perform the task and four = participant is independent in performance of task, such that overall total score may range from zero to 56 per participant. Mean Baseline and Mean Week 30 scores were calculated and used to determine change in mean score for each study group.
Time Frame: Week 30
Population: All randomized subjects are included in this analysis to determine change in mean score from Baseline to Week 30 in each study group.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Original Treatment Group: The Original Treatment Group will walk with the Ness L300 for 30 weeks.
  Ness L300: The Ness L300 delivers functional electrical stimulation (FES), which improves gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
Arm/Group | Originial Control Group | Original Treatment Group
Number analyzed (Participants) | 98 | 99
units on a scale | 3.75 (4.62) | 1.97 (6.08)
Statistical Analysis 1: Comparison: Originial Control Group vs Original Treatment Group; Test type: Superiority or Other; p < 0.022, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: User Satisfaction
Description: Total user satisfaction as measured on 12 item User Satisfaction survey with maximum score 24, minimum 0, where higher score indicated greater satisfaction with device,
Time Frame: Week 30
Population: All randomized subjects were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Originial Control Group | Original Treatment Group
Number analyzed (Participants) | 98 | 99
units on a scale | 19.1 (4.0) | 21.8 (2.9)
Statistical Analysis 1: Comparison: Originial Control Group vs Original Treatment Group; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for both study arms from Baseline to 30 weeks post-randomization.
Groups:
- Originial Control Group: The Control Group will walk with the a "usual" ankle-foot orthosis (AFO) for 30 weeks.
- Original Treatment Group: The Original Treatment Group will walk with the Ness L300 for 30 weeks.
  The Ness L300 delivers functional electrical stimulation (FES), is intended to improve gait function, stroke-specific quality of life, functionality, and safety for persons with stroke.
Arm/Group | Originial Control Group | Original Treatment Group
Serious Adverse Events (participants affected / at risk) | 7/98 | 15/99
Other Adverse Events (participants affected / at risk) | 61/98 | 82/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Originial Control Group (N=98) | Original Treatment Group (N=99)
stroke/high blood pressure (Cardiac disorders) | 1 (1) | 3 (3) — non device related
cholecystectomy (Hepatobiliary disorders) | 1 (1) | 1 (1) — non device related
pneumonia/respiratory (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — non-device related
cancer (Immune system disorders) | 1 (1) | 0 (0) — non-device related
Bone fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) — non device related
Hemiparesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — non device related
kidney damage due to dehydration (Renal and urinary disorders) | 0 (0) | 1 (1) — non device related
anemia requiring blood transfusion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — non device related
ovarian mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) — non device related
bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — non device related
methicillin resistant Staphylococcus aureus (Infections and infestations) | 0 (0) | 1 (1) — non device related
mental depression and anxiety (Psychiatric disorders) | 0 (0) | 1 (1) — non device related
hospitalization general complaints (General disorders) | 0 (0) | 1 (1) — non device related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Originial Control Group (N=98) | Original Treatment Group (N=99)
localized skin redness, rash, irritation (Skin and subcutaneous tissue disorders) | 35 (45) | 45 (68)
Eye irritation and hemorrhage (Eye disorders) | 1 (2) | 0 (0)
seasonal allergies (Immune system disorders) | 1 (1) | 0 (0)
hypertonia, headache, dizziness, memory deficit (Nervous system disorders) | 8 (9) | 8 (10)
Nausea or abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2)
Hypertension and/or flushing (Vascular disorders) | 5 (5) | 4 (4)
joint pain (Musculoskeletal and connective tissue disorders) | 21 (23) | 26 (33)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Fear or depression (Psychiatric disorders) | 1 (1) | 3 (3)
cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
gout or diabetes (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Atrial fibrillation or abnormal heartbeat (Cardiac disorders) | 1 (1) | 1 (1)
asthma, cough, bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 3 (3)
renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
blister, folliculitis (Infections and infestations) | 5 (5) | 7 (11)
fall with or without injury (Injury, poisoning and procedural complications) | 45 (71) | 56 (81)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less